CLINICAL TRIAL: NCT02285101
Title: Recombinant Human Arginase 1 (rhArg1) in Patients With Advanced Arginine Auxotrophic Solid Tumors: Dose Escalation, Safety and PK/PD
Brief Title: Recombinant Human Arginase 1 (rhArg1) in Patients With Advanced Arginine Auxotrophic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Cancer Treatment International Limited (Industry)
Collaborators: Oncotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCT-100-005
Record Dates: First submitted 2014-10-23; First posted 2014-11-06 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Melanoma; Prostate Adenocarcinoma
Keywords: arginine auxotrophic tumors; PEG-BCT-100; arginase
MeSH Terms: conditions — Melanoma | interventions — BCT-100

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): PEG-BCT-100 at 0.5 mg/kg administered as a single dose on day 1 (week 1); if not DLTs are observed, PEG-BCT- 100 will be administered at 0.5 mg/kg on days 22 (week 4) and 29 (week 5). Patients responding to treatment or with stable disease may receive 8 additional weekly administrations of PEG-BCT-100 at 0.5 mg/kg. Beyond week 13, patients responding to treatment or with stable disease may continue to receive weekly PEG-BCT-100 at 0.5 mg/kg until disease progression at the discretion of the investigator.
  Interventions: Biological: PEG-BCT-100
- Cohort 2 (Experimental): PEG-BCT-100 at 1.0 mg/kg administered as a single dose on day 1 (week 1); if not DLTs are observed, PEG-BCT- 100 will be administered at 1.0 mg/kg on days 22 (week4) and 29 (week 5). Patients responding to treatment or with stable disease may receive 8 additional weekly administrations of PEG-BCT-100 at 1.0 mg/kg. Beyond week 13, patients responding to treatment or with stable disease may continue to receive weekly PEG-BCT-100 at 1.0 mg/kg until disease progression at the discretion of the investigator.
  Interventions: Biological: PEG-BCT-100
- Cohort 3 (Experimental): PEG-BCT-100 at 1.7 mg/kg administered as a single dose on day 1 (week 1); if not DLTs are observed, PEG-BCT- 100 will be administered at 1.7 mg/kg on days 22 (week 4) and 29 (week 5). Patients responding to treatment or with stable disease may receive 8 additional weekly administrations of PEG-BCT-100 at 1.7 mg/kg. Beyond week 13, patients responding to treatment or with stable disease may continue to receive weekly PEG-BCT-100 at 1.7 mg/kg until disease progression at the discretion of the investigator.
  Interventions: Biological: PEG-BCT-100
- Cohort 4 (Experimental): PEG-BCT-100 at 1.7 mg/kg administered as a single dose on day 1 (week 1); if not DLTs are observed, PEG-BCT- 100 will be administered at 2.7 mg/kg on days 22 (week 4) and 29 (week 5). Patients responding to treatment or with stable disease may receive 8 additional weekly administrations of PEG-BCT-100 at 2.7 mg/kg. Beyond week 13, patients responding to treatment or with stable disease may continue to receive weekly PEG-BCT-100 at 2.7 mg/kg until disease progression at the discretion of the investigator.
  Interventions: Biological: PEG-BCT-100
- Cohort 5 (Experimental): PEG-BCT-100 at 1.7 mg/kg administered as a single dose on day 1 (week 1); if not DLTs are observed, PEG-BCT- 100 will be administered at 4.0 mg/kg on days 22 (week 4) and 29 (week 5). Patients responding to treatment or with stable disease may receive 8 additional weekly administrations of PEG-BCT-100 at 4.0 mg/kg. Beyond week 13, patients responding to treatment or with stable disease may continue to receive weekly PEG-BCT-100 at 4.0 mg/kg until disease progression at the discretion of the investigator.
  Interventions: Biological: PEG-BCT-100
- Cohort 6 (Experimental): PEG-BCT-100 at a dose to be determined administered as a single dose on day 1 (week 1); if not DLTs are observed, PEG-BCT-100 will be administered at at a dose to be determined on days 22 (week 4) and 29 (week 5). Patients responding to treatment or with stable disease may receive 8 additional weekly administrations of PEG-BCT-100 at at a dose to be determined. Beyond week 13, patients responding to treatment or with stable disease may continue to receive weekly PEG-BCT-100 at at a dose to be determined until disease progression at the discretion of the investigator.
  Interventions: Biological: PEG-BCT-100

INTERVENTIONS:
Biological: PEG-BCT-100
  Other Names: pegylated recombinant human arginase

SUMMARY:
The goal of this clinical research study is to evaluate the safety of PEG-BCT- 100 given as an infusion to treat patients who bear advanced solid tumors that are dependent on arginine (melanoma, renal cell carcinoma, prostate cancer and hepatocellular carcinoma), and who have progressed after receiving approved or established therapies. This is a Phase 1 study; PEG-BCT-100 is an enzyme that degrades arginine and is an investigational drug.

DETAILED DESCRIPTION:
This is a phase 1, multiple sites, open label and non-randomized study to evaluate the safety of PEG-BCT-100. Patient enrollment and sample size will follow a classical 3 + 3 dose-escalation design. The study will enroll a maximum of 36 patients. Cohorts of 3 patients will receive an initial single dose of PEG-BCT-100 beginning at 0.5 mg/kg. Single dose safety parameters including hematology and chemistry laboratory profiles will be monitored for 3 weeks. Patients not demonstrating a dose-limiting toxicity (DLT) following the single dose may then receive two additional doses of PEG-BCT-100 at the same dose level on Day 22 and Day 29. After these 2 additional doses, patients will undergo a full tumor and safety assessment after Day 29. Patients whose cancer is stable or responding may then receive weekly doses of PEG-BCT- 100 until disease progression. Dose escalations are planned for the next cohorts of 3 patients, which will be enrolled after Day 22 of the previous cohort, assuming that no single dose DLTs were reported. Each cohort of 3 patients may begin weekly administration if there is no DLTs by Day 22, and if the previous and lower dose cohort has successfully passed Week 4 of the study (doses on Days 1, and 22 + one week).

As of the beginning of 2018, an additional 22 patients will include only malignant melanoma patients. All newly enrolled patients will be enrolled at the dose level of Cohort Four (2.7 mg/kg) of PEG-BCT-100.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Stage IIIb/IV malignant melanoma or castration resistant adenocarcinoma of prostate (CRPC).
* Advanced cancer not candidate for treatment with modality or agents that are approved or have established efficacy. Candidates who cannot tolerate standard treatment or whose cancers have progressed on current standard of care.
* Males or females 18 years-old and above.
* Ability to understand and willingness to provide written informed consent;
* Karnofsky performance status (see Appendix 13.3) of 80% or above and expected survival of more than 12 weeks.
* Negative urine pregnancy test, if female, and willingness to use an effective method of contraception during the entire study period whether the patient is male or female.

Exclusion Criteria:

* Has received cancer treatment, e.g. chemotherapy, targeted biologic or enzymes, either approved or investigational, within 4 weeks prior to the start of the PEG-BCT-100;
* Advancing liver failure indicated by uncontrolled ascites, pleural effusions, or encephalopathy.
* Child-Pugh score of B and C (see Appendix 13.4).
* Significant hepatic, renal or bone marrow dysfunction indicated by: total bilirubin >2.0 mg/dL, evidence of bile duct obstruction, serum albumin <2.5 g/dL, serum ALT or AST >2.5 x upper limit of normal, serum creatinine ≥1.5 mg/dL, ANC ≥1.5 x 109/L, platelets <100 x 109/L, or INR >2.0.
* Significant cardiac or pulmonary disease defined by New York Heart Association (NYHA) Class III or IV (see Appendix 13.5), left ventricular ejection fraction (LVEF) lower than institutional normal limits by echo or MUGA, history of myocardial infarction within the past 6 months, significant unstable arrhythmia or evidence of ischemia on ECG.
* Pregnant or nursing women. NOTE: Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Significant active infection including HIV requiring oral or parenteral anti-infective therapies.
* Use of investigational drug(s) within 4 weeks of enrollment.
* Prior treatment with arginine depleting agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-11; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Number of patients undergoing adverse events (AEs) or serious adverse events (SAEs) | at least 13 weeks
Optimal Biological Dose | 13 weeks
  The optimal biological dose (OBD) of PEG-BCT-100 will be calculated based on the pharmacodynamics (PD) endpoint of plasma arginine depletion relative to plasma pharmacokinetics (PK) of PEG-BCT-100

SECONDARY OUTCOMES:
Maximum Tolerated Dose and Dosing Schedule | 4 weeks of treatment
Overall response | 13 weeks
  Evaluate objective tumor responses by RECIST (Response Evaluation Criteria In Solid Tumors)
Pharmacokinetics (PK)-PEG-BCT-100 concentration | 13 weeks
  Determine the dose-related peak to trough concentrations of plasma PEG-BCT-100 over time
Pharmacodynamics (PD) | 13 weeks
  To determine the magnitude of plasma arginine depletion (AD) relative to the dose of PEG-BCT-100
PK-PEG-BCT-100 plasma clearance | 13 weeks
  the plasma clearance of PEG-BCT-100
PD-duration of AD | 13 weeks
  the time and duration of effective AD assessed by plasma arginine <8 µM relative to the plasma peak and time to clearance over the range of PEG-BCT-100 doses
PD-relationship between AD and PEG-BCT-100 dose | 13 weeks
  the temporal and quantitative relationships of depleted plasma arginine to dose and plasma concentrations of PEG-BCT-100
PD-relationship between PEG-BCT-100 dose and tumor markers | 13 weeks
  the temporal and quantitative relationships of depleted plasma arginine to dose and plasma concentrations of PEG-BCT-100; and, The relationship of PEG-BCT-100 dose and its resultant effective AD to changes in AFP/PSA and/or tumor symptoms and measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Bessudo, MD, Principal Investigator — California Cancer Associates For Research and Excellence, cCARE; Steven O'Day, MD, Principal Investigator — Saint John's Cancer Institute
Locations (2):
- United States (2):
  - California Cancer Associates for Research and Excellence, cCARE, San Diego, California
  - John Wayne Cancer Institute, Santa Monica, California

REFERENCES:
- [Derived] De Santo C, Cheng P, Beggs A, Egan S, Bessudo A, Mussai F. Metabolic therapy with PEG-arginase induces a sustained complete remission in immunotherapy-resistant melanoma. J Hematol Oncol. 2018 May 18;11(1):68. doi: 10.1186/s13045-018-0612-6. PMID 29776373